CLINICAL TRIAL: NCT03762109
Title: The Use of Dantrolene to Improve Analgesia in Posterior Lumbar Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Richard J. Pollard, Director, Neurosurgical Anesthesia Fellowship, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018P000799
Record Dates: First submitted 2018-11-30; First posted 2018-12-03 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Lumbar Spine Injury
Keywords: Surgery; Dantrolene; Anesthesia
MeSH Terms: conditions — Spinal Injuries | interventions — Dantrolene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dantrolene Group (Experimental): Patients will receive 25 mg of Dantrolene orally at four different time points: immediately before surgery, as well as at 12, 24 and 36 hours after surgery.
  Interventions: Drug: Dantrolene
- Placebo Oral Tablet Group (Placebo Comparator): Patients will receive a 25 mg of a placebo pill orally at four different time points: immediately before surgery, as well as at 12, 24 and 36 hours after surgery.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Dantrolene — muscle relaxant
  Other Names: Dantrium; Dantrolene Sodium
  Arms: Dantrolene Group
Drug: Placebo Oral Tablet — inactive pill
  Other Names: placebo
  Arms: Placebo Oral Tablet Group

SUMMARY:
The purpose of this study is to determine whether administration of a non-centrally acting muscle relaxants will improve the Overall Benefit of Analgesia Score (OBAS), and Richmond Agitation Sedation Scale (RASS) scores in patients undergoing lumbar fusion.

ELIGIBILITY:
Inclusion Criteria

* 18 - 80 years of age (inclusive)
* Presenting to the study hospital for lumbar decompression and/or fusion (instrumented fusion of the lumbar spine < 4 levels) under general anesthesia, and scheduled for same-day admission or in-patient admission
* American Society of Anesthesiologists (ASA) Category 1, 2 or 3

Exclusion Criteria

* Known allergy to Dantrolene, morphine or other opioids, benzodiazepines that causes a reaction of hives, anaphylaxis, shock, unconsciousness/fainting, rashes/blisters, irregular heartbeat, fever, swelling, shortness of breath, wheezing, serum sickness, drug induced anemia, drug reaction with eosinophilia, and systemic symptoms, or nephritis
* Oxygen saturation < 94%
* Patient being treated with any of the following medications:Non-dihydropyridine Calcium Channel Blockers including verapamil, Estrogen therapy
* Current or past medical history of any of the following: hepatic impairment (including history of transplant), renal impairment or chronic renal disease (including history of transplant), chronic alcohol abuse, chronic respiratory disease (i.e. chronic hypoxia or hypercapnia, COPD)
* Recent history of aspiration (within the last 3 months)
* Patients with any history of neuromuscular dysfunction
* History of obstructive sleep apnea
* Weight > 140 kg
* Currently pregnant
* Actively breastfeeding
* Inability to provide written informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Overall Benefit of Analgesia Score (OBAS) | Measured at 24 hours after surgery
  OBAS scores will be recorded on a scale from 0 (best outcome) to 28 (worst outcome).

SECONDARY OUTCOMES:
Overall Benefit of Analgesia Score (OBAS) | Measured at 48 hours after surgery
  OBAS scores will be recorded on a scale from 0 (best outcome) to 28 (worst outcome).
Richmond Agitation Sedation Scale (RASS) | Measured at 24 and 48 hours after surgery
  The Richmond Agitation and Sedation Scale (RASS) is a validated and reliable method to assess patients' level of sedation in the intensive care unit. Scores range from +4 (combative) to -5 (unarousable). A score of 0 (alert and calm) is considered the best outcome.
Numerical Rating Scale (NRS) for Pain | Measured at 0, 1, 2, 3, 24, 48 hours after surgery
  Pain scores will be recorded on a scale from 0 (best outcome) to 10 (worst outcome).
ICU Length of Stay | Until discharge from the hospital, on average 24 hours
  The length of the patients stay in the ICU will be measured in hours
Hospital length of stay | Until discharge from the hospital, on average three days
  The length of the patients stay in the hospital will be measured in days
Benzodiazepine use postoperatively | Until discharge from the hospital, on average three days
  The number of patients who receive benzodiazepines after surgery will be recorded.
Morphine Equivalent Dose | Duration of the patient's stay in the hospital, on average three days
  The postoperative analgesia requirement of narcotic medications during the patients recovery will be measured in morphine equivalent dose (miligrams)
ICU Mobility Score | Measured at 24 and 48 hours after surgery
  The patients ability to move will be recorded on a scale from 0 (nothing, lying in bed; worst outcome) to 10 (walking independently without a gait aid; best outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Pollard, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No